CLINICAL TRIAL: NCT02421185
Title: A Phase 1/2a Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of JNJ-42756493, a Pan-Fibroblast Growth Factor Receptor (FGFR) Tyrosine Kinase Inhibitor, in Subjects With Advanced Hepatocellular Carcinoma
Brief Title: Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of JNJ-42756493 (Erdafitinib) in Participants With Advanced Hepatocellular Carcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR106971; 42756493HCC1001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2015-04-15; First posted 2015-04-20 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Carcinoma, Hepatocellular; JNJ 42756493; a pan-Fibroblast Growth Factor Receptor Tyrosine Kinase Inhibitor
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — erdafitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (1):
- Part 1: Dose Escalation and Part 2: Dose Expansion (Experimental): Part 1: First, participants will receive 8 milligram (mg) (starting dose) tablet of JNJ-42756493 (erdafitinib) orally once daily from Day 1 to 7, then Day 15 to 21 of 28 days cycle or 8 mg orally once daily from Day 1 to 21 of 28 days cycle (intermittent dosing). After recommended Phase 2 dose (RP2D) is identified, enrollment of continuous dosing schedule will be open, starting at 8mg. In this cohort, participants will receive 8mg (starting dose) tablet of JNJ42756493 (erdafitinib) orally once daily from Day 1 to Day 28 in a 28-day cycle. Dose of the study medication will be escalated sequentially till the dose limiting toxicity is achieved to determine RP2D.
  Part 2: Participants will receive RP2D JNJ-42756493 (erdafitinib) dose determined in Part 1. Participants who are tolerating study drug treatment and achieve clinical responses or stable disease will continue to receive study drug at the same dose until disease progression, unacceptable toxicity, or withdrawal of consent.
  Interventions: Drug: JNJ-42756493 (erdafitinib)

INTERVENTIONS:
Drug: JNJ-42756493 (erdafitinib) — Part 1: Participants will receive 8 mg tablet once daily from Day 1 to 7, and then Day 15 to 21 of 28 days cycle or 8 mg orally once daily of 28 days cycle up to the maximum tolerated dose in order to determine the recommended Phase 2 dose.
  Part 2: Recommended Phase 2 JNJ-42756493 (erdafitinib) dose determined in Part 1.

SUMMARY:
The purpose of this study is to determine recommended Phase 2 dose [RP2D]) and the objective response rate of JNJ-42756493 (erdafitinib) in advanced hepatocellular carcinoma (HCC) participants with fibroblast growth factor (FGF) 19 amplification.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), multicenter (when more than one hospital or medical school team work on a medical research study), 2 parts (First, dose escalation Phase and second, dose expansion Phase) study to evaluate the safety, pharmacokinetics, pharmacodynamics, and clinical responses of JNJ-42756493 (erdafitinib) in Asian participants with advanced HCC. The duration of study will be approximately 11 months per participant. The study consists of 2 periods: Screening (28 days before study commences on Day 1); Open-label Treatment (dose escalation portion of the trial [Part 1]), participants are enrolled into cohorts at increasing dose levels of JNJ-42756493 (erdafitinib) in 28 day treatment cycles. Part 2, the cohort expansion part of the trial, will further explore the recommended phase 2 dose (RP2D) of JNJ-42756493 (erdafitinib) as determined in Part 1; and follow-up Phase (up to 6 months). Blood samples will be collected for evaluation of safety, pharmacokinetics, pharmacodynamics, and predictive biomarkers at pre-dose and post-dose of study treatment. Recommended Phase 2 dose (RP2D) for JNJ-42756493 (erdafitinib) will be evaluated primarily. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed hepatocellular carcinoma (HCC). (histology or cytology from prior tumor biopsy specimen is acceptable). For Part 1 continuous dosing regimen and Part 2, HCC participants must have fibroblast growth factor (FGF) 19 amplification based on central laboratory results
* Participant must have advanced disease and meet all the following criteria: Disease progression after previous surgical or local-regional therapy, if any; Disease ineligible for surgical or local-regional therapy or systemic therapy; Received no more than 1 line of systemic therapy (Participants who are intolerant to previous systemic therapy are allowed.)
* Cirrhotic status of Child-Pugh class A: Participants with Child-Pugh class B score of 7 may be considered in Part 2 if no pharmacokinetic (PK) and safety issues are identified in Part 1 from subjects with Child-Pugh class A
* Eastern Cooperative Oncology Group (ECOG) performance status score 0 or 1
* Participants with adequate bone marrow, liver, renal function, and electrolytes according to protocol-defined criteria within the 14 days before the first dose of study drug
* Negative pregnancy test (urine or serum beta human chorionic gonadotropin [beta (b)-hCG]) at Screening for women of child bearing potential who are sexually active

Exclusion Criteria:

* Received systemic chemotherapy, targeted therapies, definitive radiotherapy, or treatment with an investigational anticancer agent within 2 weeks (in the case of nitrosoureas and mitomycin C, within 6 weeks; in the case of immunotherapy, within 4 weeks) before the first administration of study drug
* Prior liver transplant
* Known fibrolamellar HCC or mixed cholangiocarcinoma and HCC
* Clinically active serious infections greater than (>) Common Terminology Criteria for adverse events (AEs) grade 2
* Participants with persistent calcium or phosphate > upper limits of normal (ULN) during screening (within 14 days prior to Day 1 of Cycle 1 up until pre-dose of Cycle 1) and despite medical management of calcium or phosphate levels

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2015-05-25 (Actual); Primary Completion 2019-05-13 (Actual); Study Completion 2019-05-16 (Actual)

PRIMARY OUTCOMES:
Part 1:Recommended Phase 2 Dose (RP2D) | Up to Part 1 Day 84 (Cycle 3, Day 28) (approximately 84 days)
  RP2D will be determined based on pharmacodynamics, biomarker response or clinical response, as well as the incidence rate and nature of the toxicities observed.
Number of participants with Objective Response | up to Month 12
  Objective response based on assessment of confirmed Complete response (CR) or partial response (PR) according to modified Response Evaluation Criteria in Solid Tumors (mRECIST) for HCC. CR defined as disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to less than 10 millimeter (mm). PR defined as at least 30 percent (%) decrease in sum of the diameters of the target lesions taking as reference the Baseline sum diameters. Confirmed responses are those that persist on repeat imaging study for at least 4 weeks after initial documentation of response.

SECONDARY OUTCOMES:
Number of Participants With Adverse Events | up to Month 12
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Time to Progression (TTP) | up to Month 12
  Time interval in months between the date of randomization and the date of disease progression or death due to progression, whichever occurred first.
Disease Control Rate (DCR) | up to Month 12
  DCR defined as the proportion of participants with complete response [CR], partial response [PR], or stable disease [SD]), and duration of objective response (DOR).
Progression-free Survival | up to Month 12
  Time from date of randomization to date of first documentation of objective tumor progression or death due to any cause, whichever occurred first.
Maximum Observed Plasma Concentration of JNJ-42756493 (erdafitinib) | Up to Part 2 Day 84 (Cycle 3, Day 28) (approximately 84 days)
Time of Maximum Observed Plasma Concentration of JNJ-42756493 (erdafitinib) | Up to Part 2 Day 84 (Cycle 3, Day 28) (approximately 84 days)
Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) | Up to Part 2 Day 84 (Cycle 3, Day 28) (approximately 84 days)
  The AUCtau is the measure of the plasma drug concentration from time zero to end of dosing interval. It is used to characterize drug absorption.
Half life of JNJ-42756493 (erdafitinib) | Up to Part 2 Day 84 (Cycle 3, Day 28) (approximately 84 days)
Apparent Volume of Distribution at Steady-State of JNJ-42756493 (erdafitinib) | Up to Part 2 Day 84 (Cycle 3, Day 28) (approximately 84 days)
Total Clearance of JNJ-42756493 (erdafitinib) | Up to Part 2 Day 84 (Cycle 3, Day 28) (approximately 84 days)
Accumulation Index of JNJ-42756493 (erdafitinib) | Up to Part 2 Day 84 (Cycle 3, Day 28) (approximately 84 days)
Duration of Objective Response (DOR) | Up to Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (10):
- China (6):
  - Changchun
  - Guangzhou
  - Hangzhou
  - Harbin
  - Nanjing
  - Shanghai
- Seoul, South Korea
- Taiwan (3):
  - Kaohsiung City
  - Tainan
  - Taipei

REFERENCES:
- See also: A Phase 1/2a Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of JNJ-42756493, a pan-Fibroblast Growth Factor Receptor (FGFR) Tyrosine Kinase Inhibitor, in Subjects with Advanced Hepatocellular Carcinoma (HCC) — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CR106971&attachmentIdentifier=a83f6736-1bf3-4f4f-8db2-b6dcfbce350e&fileName=CR106971_CSR_Synopsis.pdf&versionIdentifier=